CLINICAL TRIAL: NCT00982722
Title: Vitamin D Supplementation After Successful Parathyroid Surgery for Primary Hyperparathyroidism
Brief Title: Vitamin D Supplementation After Parathyroid Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Inga-Lena Nilsson, Assoc prof, senior consultant, Karolinska University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: Eudra CT 2007-003691-19
Record Dates: First submitted 2009-09-22; First posted 2009-09-23 (Estimated); Last update posted 2019-02-28 (Actual); Status verified 2019-02

CONDITIONS: Primary Hyperparathyroidism
Keywords: primary hyperparathyroidism; postoperative vitamin D supplementation
MeSH Terms: conditions — Hyperparathyroidism, Primary | interventions — Cholecalciferol; Calcium Carbonate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- cholecalciferol and calcium carbonate (Experimental): cholecalciferol 800 IUx2 and calcium carbonate 500 mg x 2
  Interventions: Drug: calcium carbonate
- calciumcarbonate (Active Comparator): calcium carbonate 500 mg x 2
  Interventions: Drug: cholecalciferol and calcium carbonate

INTERVENTIONS:
Drug: cholecalciferol and calcium carbonate — cholecalciferol 800 IUx2 and calcium carbonate 500 mg x 2 one year after parathyroid adenomectomy, initiated 6 weeks after surgery
  Other Names: calcium carbonate
  Arms: calciumcarbonate
Drug: calcium carbonate — calcium carbonate 500 mg x 2 one year after parathyroid adenomectomy, initiated 6 weeks after surgery
  Other Names: cholecalciferol and calcium carbonate
  Arms: cholecalciferol and calcium carbonate

SUMMARY:
A randomised double blind clinical trial, accepted by the Medical Products Agency and registered in the European Clinical Trials Database. Aims to evaluate the prevalence of vitamin D deficiency in a pHPT population in relation to gender and age, the correlation between vitamin D status, pre- and postoperative parathyroid hormone level and bone density and the correlation between vitamin D status, metabolic, cardiovascular risk factors and QoL aspects before and after parathyroid adenomectomy.

DETAILED DESCRIPTION:
150 PHPT patients were randomized six weeks after surgery, 75 into each group, to 1 year of oral treatment with either calcium carbonate 1 g (500 mg twice daily) alone or calcium carbonate 1 g combined with cholecalciferol 1600 IU (800 IU twice daily). Exclusion criteria were age under 18, manifest osteoporosis at PHPTdiagnosis, persistent hypercalcemia after surgery, postoperative hypocalcemia requiring vitamin D treatment, glomerular filtration rate (GFR) below 40 ml/min, pregnancy, breast feeding, or logistical difficulties, for example living far from the hospital. Included patients had to withdraw any current supplementation with calcium and vitamin D during the study period. All tablets were identical in appearance, the tins were numbered and randomization followed a list compiled by an independent clinical research support organization. The time for randomization was chosen to make sure that the PHPT patients were cured before starting the study medication. Nearly three-quarters of the patients were randomized within 6 weeks after PTX.The primary end point was the change in PTH after PTX and treatment with the study medication. Secondary end points were vitamin D levels, insulin resistance, blood pressure and other cardiovascular risk factors, biochemical markers of bone turnover, bone mineral density and self estimated health related quality of life (SF- 36).

ELIGIBILITY:
Inclusion Criteria:

* Primary hyperparathyroidism subjected to parathyroid surgery

Exclusion Criteria:

* Renal insufficiency
* Severe osteoporosis
* Pregnancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2008-04; Primary Completion 2018-05-04 (Actual); Study Completion 2018-05-04 (Actual)

PRIMARY OUTCOMES:
postoperative parathyroid hormone level | 3 months
  PTH
ambulatory blood pressure | one year
  24h blood pressure

SECONDARY OUTCOMES:
bone mineral density | one year
  DEXA
25-OH Vitamin D | 3 months
  s-25OHD
Calcium | 6 weeks
  ionized calcium
Quality of life-self estimating formularies | one year
  SF36

CONTACTS AND LOCATIONS:
Overall Officials: Inga-Lena Nilsson, MD, Ass prof, Principal Investigator — Karolinska UH
Locations (2):
- Sweden (2):
  - Karolinska UH, Stockholm
  - Karolinska University Hospital, Stockholm

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Norenstedt S, Pernow Y, Zedenius J, Nordenstrom J, Saaf M, Granath F, Nilsson IL. Vitamin D supplementation after parathyroidectomy: effect on bone mineral density-a randomized double-blind study. J Bone Miner Res. 2014 Apr;29(4):960-7. doi: 10.1002/jbmr.2102. PMID 24115138
- [Result] Norenstedt S, Pernow Y, Brismar K, Saaf M, Ekip A, Granath F, Zedenius J, Nilsson IL. Primary hyperparathyroidism and metabolic risk factors, impact of parathyroidectomy and vitamin D supplementation, and results of a randomized double-blind study. Eur J Endocrinol. 2013 Oct 21;169(6):795-804. doi: 10.1530/EJE-13-0547. Print 2013 Dec. PMID 24026893
- [Result] Aberg V, Norenstedt S, Zedenius J, Saaf M, Nordenstrom J, Pernow Y, Nilsson IL. Health-related quality of life after successful surgery for primary hyperparathyroidism: no additive effect from vitamin D supplementation: results of a double-blind randomized study. Eur J Endocrinol. 2015 Feb;172(2):181-7. doi: 10.1530/EJE-14-0757. Epub 2014 Nov 20. PMID 25414430
- [Result] Nilsson IL, Norenstedt S, Granath F, Zedenius J, Pernow Y, Larsson TE. FGF23, metabolic risk factors, and blood pressure in patients with primary hyperparathyroidism undergoing parathyroid adenomectomy. Surgery. 2016 Jan;159(1):211-7. doi: 10.1016/j.surg.2015.06.057. Epub 2015 Oct 2. PMID 26435425
- [Result] Nilsson IL, Norenstedt S, Zedenius J, Pernow Y, Branstrom R. Primary hyperparathyroidism, hypercalciuria, and bone recovery after parathyroidectomy. Surgery. 2017 Aug;162(2):429-436. doi: 10.1016/j.surg.2017.02.017. Epub 2017 May 15. PMID 28522130